CLINICAL TRIAL: NCT02460042
Title: CONSEQUENT ALL COMERS Clinical PMCF on Peripheral Arteries Treated With SeQuent® Please OTW Paclitaxel Coated Balloon Catheter in an All Comer Patient Population
Brief Title: Clinical Post Market Clinical Follow-up (PMCF) on Peripheral Arteries Treated With SeQuent® Please Over The Wire (OTW)
Acronym: CONSEQUENT
Status: Active, not recruiting | Type: Observational
Sponsor: B. Braun Melsungen AG (Industry)
Responsible Party: Sponsor
Other Study IDs: AAG-O-H-1309
Record Dates: First submitted 2015-02-26; First posted 2015-06-02 (Estimated); Last update posted 2025-02-11 (Actual); Status verified 2025-02

CONDITIONS: Peripheral Arterial Occlusive Disease
MeSH Terms: conditions — Peripheral Arterial Occlusive Disease 1

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Procedure: drug coated balloon angioplasty — percutaneous transluminal angioplasty with peripheral balloon catheters
  Other Names: peripheral drug eluting balloon
Device: SeQuent® Please OTW Paclitaxel Coated Balloon Catheter

SUMMARY:
The aim of the study is to assess the safety and efficacy of the paclitaxel-releasing balloon catheter SeQuent® Please OTW to treat de novo and restenotic lesions in peripheral arteries. It is the intention of this trial to treat suitable target lesions with drug coated balloon (DCB) only.

DETAILED DESCRIPTION:
This study is an non-randomized, prospective, multi-center, non-interventional study (NIS=registry, for Germany: §23b MPG)

ELIGIBILITY:
Inclusion Criteria (patient):

* Willingness to treat the target lesion according to the DCB only concept
* Patients in Rutherford classes 2 through 5
* Patients eligible for peripheral revascularization by means of Percutaneous Transluminal Angioplasty (PTA)
* Patients must be 18 years of age
* Patients who are mentally and linguistically able to understand the aim of the study and to show sufficient compliance in the following study protocol
* Patients must agree to undergo at least the 12-month clinical follow-up
* Patient is able to verbally acknowledge an understanding of the associated risks, benefits, and treatment alternatives to therapeutic options of this trial, e.g. balloon angioplasty by means of the paclitaxel-eluting PTA-balloon catheter or other suitable devices. Patients, by providing their informed consent, agree to these risks and benefits as stated in the patient informed consent document.

Inclusion Criteria (lesion):

* Peripheral lesions in peripheral arteries above and below the knee with reference vessel diameters between 1.5 and 8.0 mm, lesion lengths ≥ 2 cm and ≤ 27 cm as angiographically documented*
* Diameter stenosis pre-procedure must be 70%
* Target lesion above and below the knee
* Vessels must have adequate runoff with at least one vessel to the foot. *Lesions separated by less than 2 cm are considered as one lesion

Exclusion Criteria (all comers):

* Patient not suitable for revascularization by interventional means

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with peripheral artery occlusive disease (PAOD)
Sampling Method: Probability Sample
Enrollment: 960 (Actual)
Dates: Start 2015-05 (Actual); Primary Completion 2018-12 (Actual); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Target Lesion Revascularization Rate | 12 months
  rate of target lesion revascularization (interventional, surgical)

SECONDARY OUTCOMES:
Target Lesion Revascularization Rate (TLR) | 24 months
  Target Lesion Revascularization Rate at 24 months* to establish a 'freedom from TLR' Kaplan-Meier curve
Procedural success | 1 day
  Procedural success to pass and treat the lesions (remaining stenosis is 30 %)
Ankle Brachial Index (ABI) | 12 months
  ankle brachial index
Ankle Brachial Index (ABI) | 24 months
  ankle brachial index
Ankle Brachial Index (ABI) | 3 years
  ankle brachial index
Ankle Brachial Index (ABI) | 5 years
  ankle brachial index
Maximum Walking Distance (MWD) | 12 months
  maximum walking distance under standardized conditions
Maximum Walking Distance (MWD) | 24 months
  maximum walking distance under standardized conditions
Maximum Walking Distance (MWD) | 3 years
  maximum walking distance under standardized conditions
Maximum Walking Distance (MWD) | 5 years
  maximum walking distance under standardized conditions
Patency rate | 12 months
  Patency rates as observed using non-invasive Duplex ultrasound
Patency rate | 24 months
  Patency rates as observed using non-invasive Duplex ultrasound
Patency rate | 3 years
  Patency rates as observed using non-invasive Duplex ultrasound
Patency rate | 5 years
  Patency rates as observed using non-invasive Duplex ultrasound
Rutherford classifications per group at all follow-up intervals | 12/24 months and 3/5 years
  Rutherford classifications per group at all follow-up intervals
Rutherford classification distribution change at all follow-up intervals | 12/24 months and 3/5 years
  Rutherford classification distribution change at all follow-up intervals
Amputation rate | 12/24 months and 3/5 years
  Amputation rate at 12/24 months and 3/5 years and 'freedom from amputation' Kaplan-Meier curve

CONTACTS AND LOCATIONS:
Overall Officials: Ralf Langhoff, MD, Principal Investigator — St. Gertrauden Krankenhaus, Berlin, Germany
Locations (1):
- St. Gertrauden Krankenhaus, Berlin, Germany

IPD SHARING:
Plan to Share IPD: Undecided